CLINICAL TRIAL: NCT02807688
Title: PHYSICO-DSM-VR - Physical Co-morbidity, Poor Health Behaviour and Health Promotion in Verona Patients With Functional Psychoses: a Prevalence Study and a Randomised Controlled Study
Brief Title: Physical Co-morbidity, Poor Health Behaviour and Health Promotion in Verona Patients With Functional Psychoses
Acronym: PHYSICO-DSM-VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda ULSS di Verona e Provincia (Other)
Collaborators: FONDAZIONE CARIVERONA (Unknown); Universita di Verona (Other)
Responsible Party: Principal Investigator, Lorenzo Burti, Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CE 1518
Record Dates: First submitted 2016-05-30; First posted 2016-06-21 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Psychotic Disorders; Bipolar Disorders
Keywords: health promotion; lifestyles; physical comorbidity; risk factors; behavioural change
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): "Health Promotion Intervention" package including elements of psychoeducation on healthy lifestyles and practical sessions of physical activity, with the use of motivational techniques.
  Interventions: Behavioral: Health Promotion Intervention
- Control (No Intervention): Control subjects receive treatment as usual at the Community Mental Health Services of the Department of Mental Health.

INTERVENTIONS:
Behavioral: Health Promotion Intervention — The intervention package consists of the following elements:
  i. educational sessions on the importance of diet and fitness; ii. motivational interviews to maintain participants in the program, to discuss participants' physical conditions, habits and opinions as to diet and fitness; iii. monitoring the participation in the program and health behaviour, specifically for diet and fitness, and adherence to the intervention on diet and fitness; iv. regular physical exercise under the guide and supervision of an expert trainer.
  Arms: Intervention

SUMMARY:
The study evaluates the efficacy of health promotion strategies on diet and physical activity in patients with psychosis. Half of the participants will receive an intervention protocol based on education and behavioural change, while half will not receive it.

DETAILED DESCRIPTION:
Epidemiological studies investigating the mortality and physical health of mental patients have provided substantial evidence of an excess mortality and of a substantially higher prevalence of physical co-morbidity as compared to the general population. These findings have been related to a higher prevalence of risk factors like high blood pressure, high plasma cholesterol and obesity, unhealthy lifestyles, medication side-effects.

The number of clinical trials and intervention studies in this area is still scanty and their scientific strength is relatively modest. The present research project aims at implementing preventive strategies related to dietary habits and physical exercise, and studying their efficacy with a randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 diagnosis of affective or non-affective functional psychosis (codes F20-22, F24, F25, F28-F31, F23.3, F33.3)
* one or more contacts with the CMHS in the 3 months preceding the beginning of the recruitment
* Age 18-65

Exclusion Criteria:

* moderate or severe mental handicap (learning disability)
* organic brain disorders
* lack of capacity to consent to inclusion
* subjects already involved in individual treatment related to diet and physical exercise
* subjects deemed unable or unfit to participate in the proposed physical activities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in the number of participants that comply with WHO recommendations on diet and/or exercise | baseline, month 1, month 2, month 3, month 4, month 5 and month 6
  Following the criteria proposed by World Health Organization for a healthy lifestyle: at least 5 servings of fruit/vegetables per day and at least 30 minutes of moderate physical activity per day 5 days a week. Achieving at least one more criterion than baseline at follow up is considered a success.

SECONDARY OUTCOMES:
Physical examination | baseline
  Physical examination by psychiatrist
Long term chronic disease inventory (items 2.1-2.24; MOD.ISTAT/IMF-8/B.04-05-ISTAT) | baseline
  Questionnaire assessing chronic diseases, administered by investigators
Change in blood pressure | baseline, month 1, month 2, month 3, month 4, month 5 and month 6
Change in pulses | baseline, month 1, month 2, month 3, month 4, month 5 and month 6
Change in Body Mass Index | baseline, month 1, month 2, month 3, month 4, month 5 and month 6
Change in waist circumference | baseline, month 1, month 2, month 3, month 4, month 5 and month 6
Change in glycemia | baseline and month 6
Change in haemoglobin A1C | baseline and month 6
Change in LDL cholesterol | baseline and month 6
Change in HDL cholesterol | baseline and month 6
Change in triglyceridemia | baseline and month 6
Electrocardiogram | baseline
Medication History Schedule | baseline
  Ad hoc form filled in by psychiatrist on present and previous psychopharmacological or non psychopharmacological medications taken by the participant
36 Item Short Form Health Survey | beginning and month 6
Verona Service Satisfaction Scale - European Version | beginning and month 6

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Burti, Professor, Principal Investigator — Universita di Verona
Locations (4):
- Italy (4):
  - UOC 4° Servizio Psichiatria - ULSS 20, San Bonifacio, Verona
  - UOC 1° Servizio Psichiatria - ULSS 20, Verona, Verona
  - UOC 2° Servizio Psichiatria - ULSS 20, Verona, Verona
  - UOC 3° Servizio Psichiatria - ULSS 20, Verona, Verona

IPD SHARING:
Plan to Share IPD: Undecided